CLINICAL TRIAL: NCT01175434
Title: School-Based Preventive Asthma Care Technology: A Randomized Control Trial Using a Novel Technology to Improve Adherence
Brief Title: School-Based Preventive Asthma Care Technology: A Trial Using a Novel Technology to Improve Adherence
Acronym: SB-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jill Halterman, Associate Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 32479; 1RC1HL099432-01 (NIH)
Record Dates: First submitted 2010-04-16; First posted 2010-08-04 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- School-Based Medication Group (Experimental): For children assigned to the School-Based Medication group, an asthma coordinator will send the child's primary care physician a report indicating the child's asthma symptoms, and will recommend that the child receive a preventive asthma medication at school. If the child's doctor agrees, the preventive asthma medication will be delivered to the child's school and to his/her home by a local pharmacy. The child's school nurse will begin directly observed therapy of the preventive asthma medication at school, and will routinely assess the child's asthma symptoms throughout the school year.
  Interventions: Other: School-Based Medication Delivery
- Usual Care Group (No Intervention): Children in the Usual Care group will not receive preventive medications delivered at school. These children will continue to receive all of their asthma care from their parents and primary care physicians.

INTERVENTIONS:
Other: School-Based Medication Delivery — For children assigned to the School-Based Medication group, an asthma coordinator will send the child's primary care physician a report indicating the child's asthma symptoms, and will recommend that the child receive a preventive asthma medication at school. If the child's doctor agrees, the preventive asthma medication will be delivered to the child's school and to his/her home by a local pharmacy. The child's school nurse begin directly observed therapy of the preventive asthma medication at school, and will routinely assess the child's asthma symptoms throughout the school year.
  Arms: School-Based Medication Group

SUMMARY:
The goal of this new translational project is to test the feasibility and effectiveness of implementing school-based directly observed therapy of preventive asthma medications in a real-world setting, using state-of-the-art web-based technology for systematic screening, electronic report generation, and communication between nurses, caregivers, and primary care providers. With the use of a novel method to improve adherence and subsequently reduce morbidity, the investigators hypothesize that this novel adaptation of school-based asthma care will; 1) be feasible and acceptable among this population and among school and community stakeholders, and 2) yield reduced asthma morbidity (symptom-free days, absenteeism, and emergency room / urgent care use for asthma care). The investigators anticipate that enhancing preventive healthcare for young urban children with asthma through partnerships with the schools using a novel technology will yield improved health, prevention of suffering, decreased absenteeism from school, and reduced healthcare costs.

ELIGIBILITY:
Inclusion Criteria (all 4 criteria must be met):

1. Physician-diagnosed asthma (based on parent report).
2. Persistent asthma (criteria based on NHLBI guidelines). Any 1 of the following:

   1. An average of >2 days per week with asthma symptoms
   2. >2 days per week with rescue medication use
   3. >2 days per month with nighttime symptoms
   4. ≥2 episodes of asthma during the past year that have required systemic corticosteroids
3. Age ≥3 and ≤10 years.
4. Attending school in participating Rochester City School District preschools or elementary schools.

Exclusion Criteria:

1. Inability to speak and understand English. (*Parents unable to read will be eligible, and all instruments will be given verbally.)
2. No access to a working phone for follow-up surveys (either at the subject's home or an easily accessible alternate phone number).
3. Family planning to leave the school district within fewer than 6 months.
4. The child having other significant medical conditions, including congenital heart disease, cystic fibrosis, or other chronic lung disease, that could interfere with the assessment of asthma-related measures.
5. Children in foster care or other situations in which consent cannot be obtained from a guardian.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill S. Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Univeristy of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Halterman JS, Sauer J, Fagnano M, Montes G, Fisher S, Tremblay P, Tajon R, Butz A. Working toward a sustainable system of asthma care: development of the School-Based Preventive Asthma Care Technology (SB-PACT) trial. J Asthma. 2012 May;49(4):395-400. doi: 10.3109/02770903.2012.669441. Epub 2012 Mar 28. PMID 22455402
- [Result] Halterman JS, Fagnano M, Montes G, Fisher S, Tremblay P, Tajon R, Sauer J, Butz A. The school-based preventive asthma care trial: results of a pilot study. J Pediatr. 2012 Dec;161(6):1109-15. doi: 10.1016/j.jpeds.2012.05.059. Epub 2012 Jul 10. PMID 22785264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | School-Based Medication Group | Usual Care Group
Started | 48 | 51
Completed | 48 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | School-Based Medication Group | Usual Care Group | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 51 | 99
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.48 (1.7) | 6.98 (1.8) | 7.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 25 | 32 | 57
Region of Enrollment [Number; unit: participants]
  United States | 48 | 51 | 99

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Symptom-free Days Over 14 Days; (Symptom-free Days Are Averaged Over 4 Bi-monthly Follow-ups)
Description: The primary outcome is asthma morbidity between groups. We will measure asthma morbidity by looking at the average number of symptom-free days, over 2 weeks, at each bi-monthly follow-up time point over the school year. Number of days without asthma symptoms will be reported by the child's caregiver.
Time Frame: Average number of days, over 2 weeks, throughout the school year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | School-Based Medication Group | Usual Care Group
Number analyzed (Participants) | 48 | 51
Days | 11.33 (2.6) | 10.40 (3.4)

2. Secondary Outcome: Cost Effectiveness
Description: We will evaluate the cost effectiveness to implement and sustain the web-based system in schools. We will review the cost of the intervention using three main categories of costs; programmatic costs (costs of initiating and running the program), productivity costs, and medical costs estimated at the individual child level.
Time Frame: one year
Reporting Status: Not Posted

3. Secondary Outcome: Feasibility and Acceptability
Description: We will conduct interviews with parents and school nurses to evaluate whether this new program is feasible and acceptable among this population.
Time Frame: one year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | School-Based Medication Group | Usual Care Group
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/51
Other Adverse Events (participants affected / at risk) | 0/48 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No